CLINICAL TRIAL: NCT05731726
Title: A Phase II Study to Explore the Neoadjuvant Treatment of Serplulimab Combined with CAPEOX + Celecoxib in the Treatment of Locally Advanced Rectal Cancer
Brief Title: Serplulimab Combined with CAPEOX + Celecoxib As Neoadjuvant Treatment for Locally Advanced Rectal Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Ding Ke-Feng, Professor, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASTRUM-REC01
Record Dates: First submitted 2023-02-07; First posted 2023-02-16 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-11

CONDITIONS: PMMR; MSS; MSI-L; Locally Advanced Rectal Carcinoma
Keywords: Rectal cancer; Serplulimab; Celecoxib; CAPEOX; neoadjuvant therapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Capecitabine; Oxaliplatin; Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Serplulimab+CAPEOX+celecoxib (Experimental): articipants will receive serplulimab 300 mg every 3 weeks (Q3W) concurrently with CAPEOX regimen: Oxaliplatin(130mg/m2) on day 1 of each cycle and Capecitabine, 1000mg/m2, PO, BID, day1-14, q3w and celecoxib, 200mg, PO, BID, day1-21, q3w. Treatment repeats every 3 weeks for 6-8 cycles followed by surgery (total mesorectal excision, TME).
  Interventions: Drug: Serplilumab; Drug: Capecitabine; Drug: Oxaliplatin; Drug: Celecoxib

INTERVENTIONS:
Drug: Serplilumab — Serplulimab is an innovative monoclonal antibody targeting PD-1, developed by Shanghai Henlius Biotech, Inc.
  300 mg, q3w.
  For the timing of serplulimab, there is a subgroup developed, all enrolled patients will be divided into 2 subgroups in 1:1 ratio, the fasting group and the control group. For the fasting group patients, fasting starts from 8 p.m. the day before treatment and concludes at 12 p.m. on the treatment day, water is allowed. For the control group patients, they have meals according to their habits.
  Other Names: HLX10
Drug: Capecitabine — Given PO
  Other Names: Xeloda
Drug: Oxaliplatin — Given IV
  Other Names: OHP
Drug: Celecoxib — celebrex
  Other Names: Given PO

SUMMARY:
Colorectal cancer of Mismatch Repair-proficient (pMMR)/ Microsatellite Stability (MSS) accounts for approximately 85% of all colorectal cancer patients, which might be insensitive to immunotherapy. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Chemotherapy, such as CAPEOX regimen, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Celecoxib, a COX-2 inhibitor, can improve the immune microenvironment and have a potential to synergy with immunotherapy. Chemotherapy can improve the immunogenicity of cancer cells that might enhance the efficacy of immunotherapy. The aim of this study is to explore whether chemotherapy and cyclooxygenase (COX) inhibitors combined with anti-PD-1 monoclonal antibody (mAb) could improve efficacy for resectable colorectal cancer patient with the pMMR/MSS phenotype.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent.
2. Male or female subjects ≧ 18 years ≦ 75 of age.
3. Histological or cytological documentation of adenocarcinoma of the rectum.
4. No previous any systemic anticancer therapy for rectal cancer disease.
5. The lower margin of the tumor is less than 10cm from the anus verge.
6. cT2N1-2M0, cT3N0-2M0, cT4N0-2M0 MSS with MRF(-) assessed by MRI.
7. Primary tumor can be detected by CT or MRI.
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
9. Eligible tumor tissues were identified for MSI/MMR assays.
10. Hepatitis B Surface Antigen (HBsAg) (-).
11. If HBsAg (+) , HBV-DNA must be less than 2500 copies/mL or 500 IU/mL to be enrolled.
12. Patients with HCV antibody (-) or HCV-RNA negative can be enrolled. Aspartate aminotransferase (AST) must be ≤ 3 x ULN for the lab. If HCV-RNA is positive, patients with both alanine aminotransferase (ALT) and aspartate aminotransferase (AST) performed ≤3×ULN could be enrolled. Patients infected with both hepatitis B virus and hepatitis C virus should be excluded (positive for HBsAg or HBcAb and positive for HCV antibodies).

Exclusion Criteria:

1. Patients with recurrent rectal cancer or a history of pelvic radiotherapy.
2. Patients with a history of inflammatory bowel disease.
3. Patients with acquired immunodeficiency syndrome (AIDS-related illnesses) or known human immunodeficiency virus (HIV) disease (HIV1 antibody, HIV2 antibody, HTLV1 antibody positive) should be excluded.
4. Patients who are preparing for or have previously received an organ or bone marrow transplant.
5. History of myocardial infarction, poorly controlled arrhythmias (including QTc interval ≥470 ms in women) in the 6 months prior to enrollment (QTc interval calculated by Fridericia formula).
6. According to New York College of Cardiology (NYHA) standards for Grade III-IV cardiac insufficiency or cardiac color ultrasound: left ventricular ejection fraction (LVEF) <50%.Poor hypertension control (systolic blood pressure ≥150 mmHg and/or diastolic blood pressure ≥100 mmHg), a past hypertensive crisis or hypertensive encephalopathy.
7. Poor hypertension control (systolic blood pressure ≥150 mmHg and/or diastolic blood pressure ≥100 mmHg), a past hypertensive crisis or hypertensive encephalopathy.
8. Patients had undergone major surgery within 28 days prior to enrollment. Patients with tumor biopsy or lymph node dissection biopsy were admitted. Patients undergoing enterostomy due to intestinal obstruction were admitted.
9. The patients had previously been treated with other antibodies/drugs that target immune checkpoints, such as PD-1, PD-L1, and cytotoxic T lymphocyte-associated Antigen 4 (CTLA-4).
10. Patients are participating in other clinical studies, or plan to start this study treatment less than 14 days from the end of the previous clinical study.
11. Uncontrolled tumor-related pain.
12. A known history of severe allergy to any monoclonal antibody.
13. Known to be allergic to any oxaliplatin and capecitabine ingredients.
14. Pregnant or lactating women.
15. The investigators determined that the patient had other factors that might have led to the early termination of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rates | 1 year
  Proportion of patients experiencing a pCR to perioperative PD-1 antibody

SECONDARY OUTCOMES:
Major pathological response rates | 1 year
  The proportion of patients experiencing a major pathological response to perioperative PD-1 antibody
Rate of clinical complete response rate (cCR) | 1 year
  Proportion of patients experiencing a cCR to perioperative PD-1 antibody
R0 resection rates | 1 year
  The proportion of patients achieved a complete resection with negative margin
Treatment-related adverse events. | 1 year
  Assessed by evaluation of treatment-related adverse events.
Detection of MRD | 1year
  To detect ctDNA in peripheral blood before and after treatment
single cell sequence | 1year
  Use single cell sequence to describe changes in the microenvironment of rectal cancer before and after treatment
Disease Free Survival | 3years
  Defined as the interval from enrollment to locoregional or metastatic recurrence or the appearance or a secondary colorectal cancer or death, whichever occurs first

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital School of Medicine Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No